CLINICAL TRIAL: NCT00667381
Title: Femoral Arterial Access With Ultrasound Trial
Acronym: FAUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: C. R. Bard (Industry); University of Oklahoma (Other); US Department of Veterans Affairs (U.S. Federal Agency); Long Beach Memorial Medical Center (Other)
Responsible Party: Arnold Seto, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS# 2007-5989
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-10

CONDITIONS: Vascular Access Complications; Cardiac Catheterization; Peripheral Vascular Disease
Keywords: Ultrasound guidance; Vascular access; Vascular complications
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The combination of anatomic landmarks and fluoroscopic localization of the femoral head will be used to guide femoral arterial access.
- Ultrasound (Experimental): Patients randomized to Ultrasound will have anatomic landmarks checked and real-time ultrasound guidance to aid femoral arterial access.
  Interventions: Device: Real-time Ultrasound Guidance (Site-Rite 5 or 6 machine)

INTERVENTIONS:
Device: Real-time Ultrasound Guidance (Site-Rite 5 or 6 machine) — Real-time ultrasound guidance will be used to aid in femoral artery cannulation. This will occur with a 7 MHz ultrasound probe covered with a sterile cover.
  Other Names: Site-Rite 5 or 6 ultrasound machine.
  Arms: Ultrasound

SUMMARY:
This study is designed to evaluate the routine use of vascular ultrasound as an aid for proper placement of a femoral arterial sheath during cardiac catheterization and peripheral arterial angiography.

DETAILED DESCRIPTION:
Cardiac catheterization is conventionally performed with femoral arterial access using a combination of arterial pulse palpation, anatomical landmarks, and fluoroscopic landmarks to guide needle insertion. Vascular access complications including hematoma formation, retroperitoneal bleeding, and arterial dissection are the most common types of adverse events associated with cardiac catheterization, and have been associated with insertions above and below the level of the common femoral artery. Real-time ultrasound assistance for central venous catheter placement has been proven in multiple studies to reduce complications, and has been recommended by the Agency for Healthcare Research and Quality as a "Top 11 Highly Proven" patient safety practice. This recommendation has not yet been extended to arterial access, due to a lack of studies to date. However, ultrasound assistance is licensed for and commonly utilized for arterial access, especially in difficult patients.

In a pilot study of 71 procedures performed by the lead researcher, ultrasound guidance was associated with an improved 1st pass success rate (83% vs 47%, p=0.002), reduced risk of accidental venipunctures (0% vs 25%, p=0.002), and greater overall success in common femoral artery cannulation (89% vs 69%, p=0.048) as compared with the fluoroscopic control.

This study is a multicenter prospective randomized trial to generalize the above findings with more patients studied, a larger number of operators, and across several centers. Similar to the previous study, the ultrasound will be used real-time to visualize the femoral vein, femoral artery, and needle tract as the needle is inserted, to guide the needle towards the appropriate location in the artery. The time for insertion, number of passes, complications, and position of the insertion catheter on the femoral angiogram will be analyzed in the setting of patient factors including age, body mass index, and presence of peripheral vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and over
* Patients undergoing left heart catheterization or peripheral arterial angiography from the retrograde femoral approach
* Willingness and ability to sign consent form
* Scheduled to have procedure performed by operator trained in the ultrasound technique

Exclusion Criteria:

* Access from a site other than the common femoral artery
* Nonpalpable femoral pulses
* Creatinine > 3.0 mg/dl, unless already on dialysis
* Prisoners
* Pregnant women
* Unable or refusal to sign consent form
* Patients undergoing emergent cardiac catheterization for ST segment elevation myocardial infarction or unstable acute coronary syndrome
* Equipment unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold H Seto, MD, MPA, Principal Investigator — University of California, Irvine; Morton Kern, MD, Principal Investigator — University of California, Irvine; Mazen Abu-Fadel, MD, Principal Investigator — Oklahoma Veteran's Administration Medical Center
Locations (4):
- United States (4):
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Seto AH, Abu-Fadel MS, Sparling JM, Zacharias SJ, Daly TS, Harrison AT, Suh WM, Vera JA, Aston CE, Winters RJ, Patel PM, Hennebry TA, Kern MJ. Real-time ultrasound guidance facilitates femoral arterial access and reduces vascular complications: FAUST (Femoral Arterial Access With Ultrasound Trial). JACC Cardiovasc Interv. 2010 Jul;3(7):751-8. doi: 10.1016/j.jcin.2010.04.015. PMID 20650437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2008 and February 2009, 1014 patients presenting for elective or urgent (but not emergent) cardiac or peripheral catheterization were enrolled.
Pre-assignment Details: 10 patients (6 control, 4 US) were excluded after randomization but before procedure for no longer meeting the inclusion criteria, including cancellation of the procedure, lack of a dual-trained operator, or change in access site. Baseline and procedural data were not recorded in this group, and these were not included in any analysis.
Period: Overall Study
Arm/Group | Control | Ultrasound
Started | 501 | 503
Completed | 501 | 503
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ultrasound | Total
Number analyzed (Participants) | 501 | 503 | 1004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 255 | 273 | 528
  >=65 years | 246 | 230 | 476
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.4) | 63.5 (12.4) | 63.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 132 | 267
  Male | 366 | 371 | 737
Region of Enrollment [Number; unit: participants]
  United States | 501 | 503 | 1004

OUTCOME MEASURES:

1. Primary Outcome: Participants With Successful Common Femoral Artery Cannulation, as Determined by Femoral Angiography
Description: Femoral angiography was performed in 490 control patients and 499 ultrasound patients. In 11 control and 4 ultrasound patients, femoral angiography was either not performed or was inadequate for analysis. These patients were excluded from the primary outcome analysis but included for other analyses.
  Successful common femoral artery cannulation was defined as sheath insertion above the bifurcation of the common femoral artery and below the origin of the inferior epigastric artery. Unsuccessful sheath insertion was defined as sheath insertion outside of these markers.
Time Frame: Immediately, during procedure.
Measure: Number; unit: participants
Arm/Group | Control | Ultrasound
Number analyzed (Participants) | 490 | 499
participants | 408 | 431

2. Secondary Outcome: Time to Successful Sheath Insertion.
Description: Time was measured from first fluoroscopy of the femoral head (control group), or first application of the ultrasound probe (ultrasound group), until successful sheath insertion.
  Time was not recorded for 1 control patient, and 1 ultrasound patient, these patients were excluded from this analysis but included for other analyses.
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Ultrasound
Number analyzed (Participants) | 500 | 502
seconds | 213 (194) | 185 (175)

3. Secondary Outcome: Number of Patients With Accidental Femoral Venipunctures.
Description: Number of patients with any femoral venipunctures where an insertion was not intended, i.e. excluding patients with planned right heart catheterization. Multiple accidental venipunctures were not double counted.
  Number of attempts and venipunctures were not recorded in 1 control and 1 ultrasound patient, so the denominator is 500 control patients and 502 ultrasound patients.
Time Frame: Immediate
Measure: Number; unit: participants
Arm/Group | Control | Ultrasound
Number analyzed (Participants) | 500 | 502
participants | 79 | 12

4. Secondary Outcome: Number of Participants With Vascular Complications
Description: Vascular complications were defined as vessel thrombosis, dissection, blood transfusion, hematoma > 5cm diameter, unexplained bleeding with a drop in Hgb >4 g/dL, or access site bleeding with drop in Hgb >3 g/dL.
  Outcome was assessed by chart review, and clinical or telephone followup at 30 days. Medical records were adjudicated by a blinded independent review committee.
Time Frame: Immediate and up to 1 month after procedure.
Measure: Number; unit: participants
Arm/Group | Control | Ultrasound
Number analyzed (Participants) | 501 | 503
participants | 17 | 7

5. Other Pre Specified Outcome: Number of Patients With Successful Common Femoral Artery Placement, Among Those Patients With High Femoral Artery Bifurcations
Description: Patients found to have femoral artery bifurcations occurring over the femoral head were prospectively defined as having a high femoral bifurcation. This subgroup was prespecified for analysis during the trial designed, as it was suspected that operators would have particular difficulty inserting the sheath accurately in this population.
Time Frame: At angiogram analysis
Measure: Number; unit: participants
Arm/Group | Control | Ultrasound
Number analyzed (Participants) | 159 | 149
participants | 111 | 123

ADVERSE EVENTS:
Arm/Group | Control | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/501 | 0/503
Other Adverse Events (participants affected / at risk) | 17/501 | 7/503
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=501) | Ultrasound (N=503)
Any vascular complication (Vascular disorders) | 17 (17) | 7 (7) — Any vascular complication including bleeding requiring transfusion, Hgb decrease of >3 gm/dL with known source, vessel dissection, hematoma >5cm, pseudoaneurysm, retroperitoneal hemorrhage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No